CLINICAL TRIAL: NCT01598896
Title: Combination of Dronabinol and Clonidine for Cannabis Dependence in Patients With Schizophrenia
Acronym: DCCS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: low enrollment due to limited resources
Sponsor: Mclean Hospital (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Kevin P. Hill, MD, MHS, Instructor in Psychiatry, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010P-002262; Brain and Behavior Research (Other: Brain and Behavior Research Foundation)
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Cannabis Dependence; Marijuana Dependence
Keywords: Cannabis Dependence; Marijuana Dependence; Cannabis Use Disorders; Cannabis Withdrawal; Dronabinol; Clonidine; Schizophrenia
MeSH Terms: conditions — Marijuana Abuse; Schizophrenia | interventions — Dronabinol; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dronabinol + Clonidine (Experimental): Dronabinol titrated to 5 mg three times daily, Clonidine 0.1 mg twice daily
  Interventions: Drug: Dronabinol; Drug: Clonidine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol titrated to 5 mg three times daily
  Other Names: Marinol, CSA Drug Code 7369, Schedule III, NDC 54868-3189-0
  Arms: Dronabinol + Clonidine
Drug: Clonidine — Clonidine 0.1 mg twice daily
  Other Names: Catapres, NDC 16590-266-30
  Arms: Dronabinol + Clonidine
Drug: Placebo — One placebo capsule by mouth twice daily
  Arms: Placebo

SUMMARY:
Cannabis use disorders are an important public health problem in the United States, but no effective pharmacotherapies are available to treat these disorders. People with schizophrenia are more likely than healthy people to abuse cannabis. Cannabis use may worsen clinical outcomes in this group, making the identification of pharmacotherapy to treat cannabis dependence in those with schizophrenia important. The investigators intend to test the combination of dronabinol, a cannabinoid agonist, and the α2-adrenergic agonist clonidine, for cannabis dependence in subjects with schizophrenia. The combination of dronabinol and clonidine may alleviate cannabis withdrawal symptoms while allowing treatment-seeking outpatients to benefit from medical management (MM) sessions when they are trying to stop using cannabis. The investigators propose to assess the relationship of dronabinol and clonidine, when added to MM, on cannabis use patterns in cannabis-dependent patients with schizophrenia.

Hypothesis: The investigators predict that combination pharmacotherapy of dronabinol and clonidine will significantly reduce cannabis use compared to those receiving placebo.

DETAILED DESCRIPTION:
Subjects will receive either the combination of dronabinol and clonidine or placebo in addition to medical management (MM) over a 10-week treatment period. Following treatment completion, subjects will have follow-up visits until 14 weeks after treatment initiation. This pilot study will evaluate the feasibility of the combination of dronabinol and clonidine for cannabis dependence and will establish effect sizes for a larger trial.

Cannabis use disorders are highly prevalent in the United States and rising among high school seniors, making the identification of efficacious treatments for cannabis dependence of critical clinical and public health significance. Schizophrenia is overrepresented among those with cannabis dependence. At the completion of this study, the investigators hope to have improved our understanding of the relationship of the pharmacotherapy combination of dronabinol and clondine on cannabis use.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-45 years
2. DSM-IV diagnosis of cannabis dependence, based on the Structured Clinical Interview for DSM-IV (SCID)
3. DSM-IV diagnosis of schizophrenia or schizoaffective disorder, based on the Structured Clinical Interview for DSM-IV (SCID)
4. express a desire to quit cannabis use within the next 30 days
5. have used cannabis on ≥20 days within the past 30 days (i.e., an average of ≥5 day per week)
6. identify cannabis as their primary drug of abuse; 6) stable on antipsychotic medication for ≥1 month
7. for women of childbearing age, a negative pregnancy test at screening with agreement to use adequate contraception to prevent pregnancy and monthly pregnancy tests
8. consent for us to communicate with their prescribing clinician if one exists
9. furnish the names of 2 locators, who would assist study staff in locating them during the study period
10. live close enough to McLean Hospital to attend study visits
11. plan to stay in the Boston area for the next 3 months
12. are willing and able to sign informed consent.

Exclusion Criteria:

1. Current diagnosis of other drug or alcohol dependence (excluding nicotine)
2. significant cardiac disease as indicated by history or suspected by abnormal ECG or history of cardiac symptoms
3. Positive and Negative Syndrome Scale (PANSS) subscale for positive symptoms of psychosis item > 3 (moderate) at baseline evaluation
4. current medical condition that could prevent regular study attendance
5. liver function tests >3 times the upper limit of normal range
6. history of seizure disorder or history of head trauma or CNS insult that could predispose the subject to seizures
7. taking clozapine
8. current suicidal risk
9. bradycardia less than or equal to 50 bpm, supine blood pressure of less than or equal to 100/65, a seated blood pressure of less than or equal to 90/60, or orthostatic change of >20 systolic or >10 diastolic on standing, at screening or any pre-dose assessment, or symptoms attributable to low BP (i.e. lightheadedness or dizziness on standing)
10. mental retardation or organic mental disorder
11. currently in a residential treatment setting in which substance use is monitored and restricted, since the restricted access to drugs could represent an important confounding variable
12. pregnant, nursing, or, if a woman of childbearing potential, not using a form of birth control judged by the investigator to be effective
13. concomitant treatment with opioid analgesics, sedative hypnotics, or other known CNS depressants
14. known hypersensitivity to cannabinoids or sesame oil or clonidine
15. disease of the gastrointestinal system, liver, or kidneys that may impede metabolism or excretion of dronabinol
16. inability to read or write in English that would hinder their ability to follow study procedures
17. history of seizures or a family history of seizures.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin P Hill, MD, MHS, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7 subjects were randomized for this study out of 12 subjects who were screened for this DCCS study at McLean Hospital
Pre-assignment Details: 5 subjects that were screened were not randomized. 1 subject stopped using MJ between the screening visit and baseline visit and was thus withdrawn, 2 subjects were no longer interested in the study after screening visit, 1 subject entered in-patient treatment before randomization and 1 screened subject did not meet DSM criteria for MJ dependence
Groups:
- Dronabinol-Clonidine: Dronabinol titrated to 5 mg three times daily
  Dronabinol: Dronabinol titrated to 5 mg three times daily
  Clonidine 0.1 mg twice daily
  Clonidine: Clonidine 0.1 mg twice daily
Period: Overall Study
Arm/Group | Dronabinol-Clonidine | Placebo
Started | 3 | 4
Completed | 3 | 2
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol + Clonidine | Placebo | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.67 (13.58) | 30.75 (5.91) | 32.86 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Self-Report MJ Use [Mean (Standard Deviation); unit: hits/day] | 37.16 (21.92) | 37.4 (19.32) | 37.3 (18.63)
Marijuana Craving [Mean (Standard Deviation); unit: Score on MCQ 4 Factor Total scale] — The baseline Marijuana Craving Questionnaire (Heishman et al. 2009) - The 4 Factor Total Score
  Maximum Score = 84 Minimum Score = 12 The higher the score, the more severe marijuana craving symptoms endorsed by the subject.
  Score on MCQ 4 Factor Total scale | 65 (10.15) | 55.5 (13.33) | 59.57 (12.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cannabis Use at 10 Weeks
Description: Subject self-report hits of marijuana per day at week 10
Time Frame: At 10 weeks
Population: Only 2 of the 4 placebo subjects had Week 10 data due to dropping out of the study.
Measure: Mean (Standard Deviation); unit: hits/day
Arm/Group | Dronabinol + Clonidine | Placebo
Number analyzed (Participants) | 3 | 2
hits/day | 16.91 (14.57) | 22.35 (17.47)

2. Secondary Outcome: Change in Craving Symptoms From Baseline at 10 Weeks
Description: Scores on the Marijuana Craving Questionnaire (MCQ) (Heishman et al. 2009) - The 4 Factor Total Score.
  Maximum Score = 84 Minimum Score = 12 The higher the score, the more severe marijuana craving symptoms endorsed by the subject.
Time Frame: At 10 weeks
Population: Only 2 of the placebo subjects completed week 10 and had MCQ scores for Week 10.
Measure: Mean (Standard Deviation); unit: score on a MCQ 4 Factor Total scale
Arm/Group | Dronabinol + Clonidine | Placebo
Number analyzed (Participants) | 3 | 2
score on a MCQ 4 Factor Total scale | 51 (15.71) | 52.33 (15.04)

3. Secondary Outcome: Change From Baseline in Cannabis Use at 14 Weeks
Description: Self-report cannabis use at 14 weeks after initiating the study.
Time Frame: At 14 weeks
Population: Only 1 of the placebo subjects had week 14 data due to the other week 10 completer not attending the follow-up visit at week 14.
Measure: Mean (Standard Deviation); unit: hits/day
Arm/Group | Dronabinol + Clonidine | Placebo
Number analyzed (Participants) | 3 | 1
hits/day | 18.95 (6.69) | 16.29 (0)

4. Secondary Outcome: Change in Craving Symptoms From Baseline at 14 Weeks
Description: Scores on the Marijuana Craving Questionnaire (Heishman et al. 2009) - The 4 Factor Total Score
  Maximum Score = 84 Minimum Score = 12 The higher the score, the more severe marijuana craving symptoms endorsed by the subject.
Time Frame: At 14 weeks
Population: Only 1 placebo subject completed Week 14 of the study and had Week 14 MCQ Total Score data.
Measure: Mean (Standard Deviation); unit: score on MCQ Total 4 Factor scale
Arm/Group | Dronabinol + Clonidine | Placebo
Number analyzed (Participants) | 3 | 1
score on MCQ Total 4 Factor scale | 54.33 (9.29) | 56 (0)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected every visit starting with the baseline visits up until the last visit of the study 14 weeks later.
Arm/Group | Dronabinol + Clonidine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol + Clonidine (N=3) | Placebo (N=4)
Nausea associated with Placebo (General disorders) | 0 (0) | 1 (1) — 1 subject called study staff to say the medication was making her nauseous. When subject was called back, the nausea was gone and did not occur again. The PI called the subject who stated it must have been unrelated to study

LIMITATIONS AND CAVEATS:
Due to lack of sufficient funds/resources, the sample size for this study is not large enough to extract any conclusive results. The high number of subjects withdrawing from the study early also hinders any possible conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT01598896/Prot_SAP_001.pdf